CLINICAL TRIAL: NCT06127186
Title: Phenotype of Headache and Facial Pain in Upper Respiratory Tract Infections - a Cross-sectional Study in Primary Care Setting
Brief Title: Phenotype of Headache and Facial Pain in Upper Respiratory Tract Infections
Status: Completed | Type: Observational
Sponsor: Marcin Straburzynski (Other)
Responsible Party: Sponsor-Investigator, Marcin Straburzynski, Principal Investigator, Swiat Zdrowia
Organization: Swiat Zdrowia (Other)
Other Study IDs: URTI HA FP
Record Dates: First submitted 2023-11-04; First posted 2023-11-13 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Upper Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients reporting for primary care assessment because of URTI.
  Interventions: Diagnostic Test: Swab test for viral antigens

INTERVENTIONS:
Diagnostic Test: Swab test for viral antigens — No intervention except for a routine examination and viral testing is planned.
  Other Names: Standarised questionnaire; Physical examination

SUMMARY:
The goal of this longitudinal study is to assess headache and facial pain features in patients with upper respiratory tract infections (URTI). The main question it aims to answer are:

1. What is the phenotype of headache / facial pain in URTIs
2. Does the above mentioned phenotype is associated with:

   1. aetiologic factor (virus),
   2. type of URTI
   3. headache/facial pain experienced by patients in the past.

Participants will:

* answer standardized questions,
* undergo physical examination,
* have a swab test performend for antigens of common viruses causing URTI.

ELIGIBILITY:
Inclusion Criteria:

* URTI confirmed by primary care physician
* Informed consent to participate in the study

Exclusion Criteria:

* chronic or recurrent upper respiratory tract disorders
* neoplasms
* signs or symptoms of a serious neurologic or psychiatric disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with upper respiratory tract infection.
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with one of the specified pain phenotypes | A single assessment during primary care physician office 1 day visit.
  Percentage of patients with one of the specified pain phenotypes (migraine-like/tension-type-like/trigeminal cephalalgia-like)

CONTACTS AND LOCATIONS:
Locations (1):
- Marcin Straburzyński, Dźwierzuty, Warmian-Masurian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be made available in a public repository after study completion.
Supporting Information: Study Protocol